CLINICAL TRIAL: NCT05118464
Title: Evaluation of the Effect of Dual-Task Training on Muscle Strength, Balance, and Gait in Pediatric Oncology Patients
Brief Title: Effect of Dual-Task Training on Pediatric Oncology Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Emel Taşvuran Horata, PhD; Assistant Professor, Afyonkarahisar Health Sciences University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020/387
Record Dates: First submitted 2021-10-31; First posted 2021-11-12 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: Cancer
Keywords: cancer; gait; postural balance; muscle strength
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children with cancer (Experimental): The arm of the research will consist of pediatric patients aged 6-18 years who have been diagnosed with cancer in Afyonkarahisar Health Sciences University, Health Application and Research Center, Department of Pediatric Hematology-Oncology Clinics and who come for outpatient treatment.
  Interventions: Other: Dual-task training

INTERVENTIONS:
Other: Dual-task training — Dual-task training includes simultaneous execution of motor and cognitive tasks. The motor tasks in this study will be walking, going up and downstairs, turning, throwing, and holding a ball. Cognitive tasks will be an n-back test, verbal fluency, remembering sequences of numbers, and performing simple summing.

SUMMARY:
It is known that the treatment of children with cancer has negative effects on cognition, muscle strength, balance, and gait. Therefore, the aim of this study is to evaluate the effects of dual-task training, which is based on the principle of simultaneous performance of cognitive tasks and motor tasks, on muscle strength, balance, and gait.

DETAILED DESCRIPTION:
With the increase in the incidence of cancer, the number of children who survived cancer is also increasing. Most studies on cancer survivors show that the disease and its treatment have side effects and long-term late effects on the musculoskeletal system, physical function, motor, and cognitive skills. Therefore, the aim of this study is to evaluate the effects of dual-task training, which is based on the principle of simultaneous performance of cognitive tasks and motor tasks, on muscle strength, balance, and gait. This study is planned to be the first study in which dual-task training is applied in children with cancer.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with pediatric cancer and inpatient and outpatient treatment in Hematology-Oncology Clinics for treatment,
* Able to walk alone without any walking aid,
* Children aged 6-18 will be included

Exclusion Criteria:

* Staying in an isolated room or at risk of infection (neutropenic, etc.),
* Any orthopedic or neurological disorder that may prevent walking;
* Having any mental disability that will prevent performing a cognitive task,
* Individuals with malignant hypertension or unstable heart disease (eg, congestive heart failure) will not be included in the study.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Estimated)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-09-15 (Estimated); Study Completion 2023-09-15 (Estimated)

PRIMARY OUTCOMES:
gait speed | 600 seconds
  Gait speed is the time one takes to walk a specified distance on level surfaces over a short distance. It will be recorded in m/s.
balance | 300 seconds
  Balance is evaluated with Timed-up and Go Test. The time elapsed during the test is recorded in seconds.
Muscle strength | 600 seconds
  Isometric muscle strength will be evaluated with a hand-held dynamometer. It will be recorded in kg.

CONTACTS AND LOCATIONS:
Overall Officials: EMEL TAŞVURAN HORATA, PhD, Principal Investigator — AFSU
Locations (1):
- Emel Taşvuran Horata, Afyonkarahisar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No